CLINICAL TRIAL: NCT01054196
Title: Lenalidomide Plus Melphalan as a Preparative Regimen for Autologous Stem Cell Transplantation in Relapsed Multiple Myeloma: A Phase 1 / 2 Study
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0909010623
Record Dates: First submitted 2010-01-19; First posted 2010-01-22 (Estimated); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1 Dose level 1 (Experimental): Oral lenalidomide 25mg twice daily x 5 days (designated as days -5 to -1).
  On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  Interventions: Drug: lenalidomide; Drug: melphalan
- Phase 1 Dose level 2 (Experimental): Oral lenalidomide 25mg qAM, 50mq qPM x 5 days (designated as days -5 to -1).
  On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  Interventions: Drug: lenalidomide; Drug: melphalan
- Phase 1 Dose level 3 (Experimental): Oral lenalidomide 50mg qAM, 75mg qPM x 5 days (designated as days -5 to -1).
  On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  Interventions: Drug: lenalidomide; Drug: melphalan
- Phase 1 Dose level 4 (Experimental): Oral lenalidomide 75mg qAM, 100mg qPM x 5 days (designated as days -5 to -1).
  On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  Interventions: Drug: lenalidomide; Drug: melphalan
- Phase 1 Dose level 5 (Experimental): Oral lenalidomide 100mg qAM, 150mg qPM x 5 days (designated as days -5 to -1).
  On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  Interventions: Drug: lenalidomide; Drug: melphalan
- Phase 1 Dose level 6 (Experimental): Oral lenalidomide 150mg qAM, 200mg qPM x 5 days (designated as days -5 to -1).
  On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  Interventions: Drug: lenalidomide; Drug: melphalan
- Phase 2 Expansion (Experimental): Early studies noted a dose response relationship and found myelosuppression to be the dose limiting toxicity. In this Phase 1 study of high dose lenalidomide (HDLEN) with HDM in conditioning for ASCT shown no DLT noted up to 350mg PO daily of LEN.
  In Phase 2, HDLEN was dosed at 350mg PO daily from day -5 to day -1 and HDM was dosed 100mg/m2 on days -2 and -1.
  After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  lenalidomide: daily dose dependent on dose-escalation schedule
  melphalan: 100 mg/m2 given Days -2 and -1
  Interventions: Drug: lenalidomide; Drug: melphalan

INTERVENTIONS:
Drug: lenalidomide — daily dose dependent on dose-escalation schedule
  Other Names: Revlimid
Drug: melphalan — 100 mg/m2 given Days -2 and -1

SUMMARY:
A) Phase 1: To determine the maximal tolerated dose (MTD) of lenalidomide that can be safely added to high-dose melphalan prior to autologous stem cell transplantation (ASCT).

B) Phase 2: To determine whether the addition of high-dose lenalidomide to ASCT followed by maintenance standard-dose lenalidomide improves the response rate and duration of response for relapsed multiple myeloma (RMM).

DETAILED DESCRIPTION:
Experimental: Phase 1 Subjects will dose escalate lenalidomide in a series of subjects in a 3+3 design through 6 dose levels of lenalidomide (as per modified Fibonacci escalation) to determine the maximal tolerated dose (MTD)of lenalidomide prior to ASCT.

Planned dose levels of lenalidomide in Phase 1 portion of study:

Dose Level/ Lenalidomide Dose / Schedule

-1: 25mg daily x 5 days

1. 25mg twice daily x 5 days
2. 25mg qAM, 50mq qPM x 5 days
3. 50mg qAM, 75mg qPM x 5 days
4. 75mg qAM, 100mg qPM x 5 days
5. 100mg qAM, 150mg qPM x 5 days
6. 150mg qAM, 200mg qPM x 5 days

Experimental: Phase 2 The MTD determine for lenalidomide in the phase 1 portion of this study will be used in the transplant phase of the phase 2 portion.

In the transplant phase of the study, all participants will receive oral lenalidomide at the pre-determined dose level for phase 1 and MTD for phase 2 for 5 days (designated as days -5 to -1). On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.

Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed relapsed, primary refractory, or relapsed and refractory multiple myeloma.
* Patients must have measurable disease as defined by the International Uniform Response Criteria,defined as any of the following:

  * serum M-protein of > = 500mg/dL
  * urine M-protein of > = 200mg/ 24 hours
  * involved free light chain > = 10mg/dL provided serum free light chain ratio is abnormal
* Patients must have received at least one prior line of therapy.
* Age > = 18 years.
* Life expectancy of greater than 12 weeks.
* ECOG performance status < = 2.
* All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist.
* Patients must have normal organ and marrow function as defined below:

  * ANC > = 1,000/uL
  * platelets > = 50,000/uL
  * total bilirubin < = 1.5 X upper limit of normal
  * AST(SGOT)/ALT(SGPT) < = 2.5 X upper limit of normal
  * Cardiac Ejection Fraction > = 45 %
  * Creatinine clearance > 60 cc/min
* Patients must have an adequate number of CD34+ stem cells collected to allow for transplantation. This number is defined as ≥ 2 x 106 CD34+ cells / kg body weight. If not previously collected and stored, the patient must be willing to undergo stem cell mobilization and collection as per standard practice.
* The effects of lenalidomide on the developing human fetus at the recommended therapeutic dose are unknown; however, it has been shown to be teratogenic other primates. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. The treating physician will follow the adverse reporting guidelines as outlined in further detail below for pregnancies.
* Lenalidomide has been shown to carry a risk of thromboembolic events, especially when used in combination with either corticosteroids or alkylating chemotherapeutic agents. All patients who participate in this study must be willing and able to tolerate prophylactic anticoagulation with low-molecular weight heparin (LMWH) for the required dates in treatment protocol. Patients also must be able to tolerate low-dose aspirin, 81 mg daily, during the maintenance phase of the treatment protocol.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had myeloma therapy within 14 days prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier. Patients may have received bisphosphonate therapy as part of routine myeloma care at any time prior to study entry.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lenalidomide (including thalidomide) or melphalan.
* Known positive for HIV or infectious hepatitis, type B or C.
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and lactating women are excluded from the study because the risks to an unborn fetus or potential risks in nursing infants are unknown.
* History of thrombosis or thromboembolic event within last 60 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Pearse, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- See also: Related Info — https://weillcornell.org/myeloma

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Level 1: Oral lenalidomide 25mg twice daily x 5 days (designated as days -5 to -1).
  On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  lenalidomide: daily dose dependent on dose-escalation schedule
  melphalan: 100 mg/m2 given Days -2 and -1
- Phase 1 Dose Level 2: Oral lenalidomide 25mg qAM, 50mq qPM x 5 days (designated as days -5 to -1).
  On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  lenalidomide: daily dose dependent on dose-escalation schedule
  melphalan: 100 mg/m2 given Days -2 and -1
- Phase 1 Dose Level 3: Oral lenalidomide 50mg qAM, 75mg qPM x 5 days (designated as days -5 to -1).
  On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  lenalidomide: daily dose dependent on dose-escalation schedule
  melphalan: 100 mg/m2 given Days -2 and -1
- Phase 1 Dose Level 4: Oral lenalidomide 75mg qAM, 100mg qPM x 5 days (designated as days -5 to -1).
  On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  lenalidomide: daily dose dependent on dose-escalation schedule
  melphalan: 100 mg/m2 given Days -2 and -1
- Phase 1 Dose Level 5: Oral lenalidomide 100mg qAM, 150mg qPM x 5 days (designated as days -5 to -1).
  On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  lenalidomide: daily dose dependent on dose-escalation schedule
  melphalan: 100 mg/m2 given Days -2 and -1
- Phase 1 Dose Level 6: Oral lenalidomide 150mg qAM, 200mg qPM x 5 days (designated as days -5 to -1).
  On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  lenalidomide: daily dose dependent on dose-escalation schedule
  melphalan: 100 mg/m2 given Days -2 and -1
Period: Overall Study
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4 | Phase 1 Dose Level 5 | Phase 1 Dose Level 6 | Phase 2 Expansion
Started | 2 | 4 | 3 | 4 | 6 | 3 | 30
Completed | 2 | 4 | 3 | 3 | 6 | 3 | 29
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase 2 MTD: Phase 2 MTD, oral lenalidomide 150mg qAM, 200mg qPM x 5 days (designated as days -5 to -1).
  On days-2 and -1, all patients will receive 100mg/m2 of intravenous melphalan once daily for a total of 2 doses (200mg/m2total). After a period of 24-72 hours has elapsed from the last melphalan dose (designated as Day 0) each patient will receive infusion of at least 2.0 x 106/kg of autologous CD34+ stem cells.
  Maintenance lenalidomide will begin at Day +100 at a dose of 25 mg/day, orally for 1-21 days followed by a 7-day rest period (28 day cycles).
  lenalidomide: daily dose dependent on dose-escalation schedule
  melphalan: 100 mg/m2 given Days -2 and -1
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4 | Phase 1 Dose Level 5 | Phase 1 Dose Level 6 | Phase 2 MTD | Total
Number analyzed (Participants) | 2 | 4 | 3 | 4 | 6 | 3 | 30 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 2 | 1 | 5 | 2 | 19 | 34
  >=65 years | 0 | 1 | 1 | 3 | 1 | 1 | 11 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 3 | 0 | 12 | 22
  Male | 1 | 2 | 1 | 2 | 3 | 3 | 18 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 0 | 0 | 5 | 7
  White | 0 | 3 | 1 | 3 | 5 | 3 | 17 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 1 | 1 | 0 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 3 | 4 | 6 | 3 | 30 | 52
Immunoglobulin Isotype [Count of Participants; unit: Participants]
  IgG Lambda | 1 | 1 | 0 | 2 | 1 | 0 | 7 | 12
  IgG Kappa | 1 | 1 | 0 | 0 | 2 | 0 | 12 | 16
  IgA Lambda | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 5
  IgA Kappa | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 6
  IgD Kappa | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Kappa Free light Chain | 0 | 1 | 2 | 0 | 3 | 1 | 3 | 10
  Lambda Free light Chain | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Lenalidomide That Can be Added to Melphalan
Description: The primary endpoint for the phase 1 portion of this study is to determine the maximum tolerated dose of lenalidomide that can be added to melphalan.
Time Frame: 12 months
Population: This outcome measure only assesses Phase 1 participants
Measure: Number; unit: mg/day
Groups:
- All Phase 1 Participants: All participants who received lenalidomide at
  25mg daily x 5 days 25mg twice daily x 5 days 25mg qAM, 50mq qPM x 5 days 50mg qAM, 75mg qPM x 5 days 75mg qAM, 100mg qPM x 5 days 100mg qAM, 150mg qPM x 5 days 150mg qAM, 200mg qPM x 5 days
Arm/Group | All Phase 1 Participants
Number analyzed (Participants) | 21
mg/day | NA — Despite administering HDLEN at doses of up to 350 mg/day, the maximum tolerated dose could not be determined, owing to an insufficient number of dose-limiting toxicities in the 21 patients enrolled in the trial

2. Primary Outcome: Duration of Overall Response (DoR)
Description: The primary endpoint for the phase 2 portion of this study is to determine the duration of overall response (DoR). The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: Until disease progression, death, or for a maximum of 3 years, whichever occurs first
Population: This outcome measure only assesses Phase 2 participants
Measure: Number; unit: participants
Arm/Group | Phase 2 Expansion
Number analyzed (Participants) | 28
participants
  sCR | 7
  CR | 6
  VGPR | 10
  PR | 4
  SD | 1
  PD | 0

3. Secondary Outcome: Overall Response Rate
Description: Overall response rate is the number of patients with complete response and partial response. Response is defined by the International Uniform Response Criteria for Multiple Myeloma (IURC)
Time Frame: Until disease progression or a maximum of 3 years, whichever occurs first
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the interval between the day of transplantation (Day 0) and date of death. If the date of death is uncertain, the date of last contact with the subject will be used.
Time Frame: Until death or date of last contact with the subject
Reporting Status: Not Posted

5. Secondary Outcome: Mean Functional Assessment of of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) Score
Description: quality of life will be evaluated and scored using the questionnaire from the bone marrow transplant subscale of the Functional Assessment of Cancer Therapy available from w ww.facit.org. The FACT-BMT is a 50 item questionnaire that measures five dimensions of quality of life in bone marrow transplant patients, including physical well-being, social and family well-being, emotional well-being, functional well-being, and additional concerns. It is scored on a 5 point Likert scale. Total scores range from 0 to 148, with a higher score indicating higher quality of life.
Time Frame: Cycle 6, day 1, at approximately 4.5 months
Population: Subjects from whom data were not collected were excluded from analysis.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4 | Phase 1 Dose Level 5 | Phase 1 Dose Level 6 | Phase 2 Expansion
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 6 | 3 | 21
score on a scale | 85.28 [0 to 148] | 69.3 [0 to 148] | 81.5 [0 to 148] | 70.13 [0 to 148] | 80.14 [0 to 148] | 79.33 [0 to 148] | 74.68 [0 to 148]

ADVERSE EVENTS:
Time Frame: Adverse events presented were collected for an average of 3 years
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4 | Phase 1 Dose Level 5 | Phase 1 Dose Level 6 | Phase 2 MTD
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/3 | 0/4 | 0/6 | 0/3 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/4 | 1/3 | 2/4 | 3/6 | 1/3 | 8/30
Other Adverse Events (participants affected / at risk) | 1/2 | 4/4 | 3/3 | 3/4 | 6/6 | 3/3 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=2) | Phase 1 Dose Level 2 (N=4) | Phase 1 Dose Level 3 (N=3) | Phase 1 Dose Level 4 (N=4) | Phase 1 Dose Level 5 (N=6) | Phase 1 Dose Level 6 (N=3) | Phase 2 MTD (N=30)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Hip pain
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Diverticulitis
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Gastroenteritis
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Umbilical abscess
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Myocardiac Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Basal cell carcinoma, lip
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=2) | Phase 1 Dose Level 2 (N=4) | Phase 1 Dose Level 3 (N=3) | Phase 1 Dose Level 4 (N=4) | Phase 1 Dose Level 5 (N=6) | Phase 1 Dose Level 6 (N=3) | Phase 2 MTD (N=30)
Abdominal Distention (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 4 (5) | 2 (3) | 1 (1)
Activated PTT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 11 (11)
Acute kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (3) | 3 (3) | 1 (1) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 20 (50)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (13) | 0 (0) | 0 (0) | 16 (35)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Acute otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (8) | 3 (4) | 3 (4) | 6 (8) | 3 (6) | 28 (59)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 4 (5) | 3 (3) | 2 (2) | 6 (6) | 3 (3) | 19 (23)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (4) | 1 (4) | 2 (2) | 2 (2) | 11 (13)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 18 (46)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (13) | 2 (2) | 1 (1) | 14 (20)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 29 (96) — Leukopenia
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 1 (2) | 10 (20)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (4) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) — eGFR decreased
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concentration impairement (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (4) | 4 (6) | 2 (4) | 8 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 7 (8)
CPK increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Creatinine increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 8 (13)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (9) | 3 (6) | 3 (17) | 6 (12) | 3 (5) | 25 (53)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 4 (5) | 2 (2) | 5 (5)
Dry eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 3 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 2 (2) | 2 (4) | 3 (3) | 2 (2) | 7 (7)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 8 (9)
Edema limb (General disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Hordeolum
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 4 (7) | 3 (3) | 3 (14) | 5 (8) | 3 (5) | 23 (38)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (4) | 3 (3) | 2 (2) | 6 (6) | 2 (3) | 7 (7)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 7 (7)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gait alteration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3)
Gastroesophageal reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 5 (5) — Odynophagia
Gastropharesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 5 (7)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hypercalcemia (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 3 (4) | 3 (8) | 3 (5) | 5 (6) | 3 (4) | 29 (68)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 4 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (9)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (8)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (11)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 27 (50)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (4) | 4 (10) | 3 (7) | 3 (10) | 6 (12) | 3 (3) | 28 (84)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (5) | 3 (10) | 3 (7) | 3 (20) | 1 (4) | 0 (0) | 15 (24)
Hypokalemia (Metabolism and nutrition disorders) | 1 (5) | 4 (6) | 3 (3) | 3 (4) | 4 (7) | 1 (1) | 25 (32)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (6) | 2 (5) | 3 (6) | 3 (18) | 5 (9) | 3 (6) | 21 (62)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 13 (21)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 2 (3) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 3 (3)
Infusion-Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INR increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 21 (28)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (10) | 3 (3) | 0 (0) | 12 (24)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (18) | 0 (0) | 0 (0) | 29 (75)
Lymphocyte count increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 2 (2) | 1 (1) | 3 (3)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (8) | 2 (4) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (7) | 3 (3) | 0 (0) | 5 (6) | 2 (2) | 21 (38)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (6) | 4 (15) | 3 (10) | 3 (18) | 6 (26) | 3 (9) | 29 (113)
Non-cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 1 (2) | 0 (0) | 17 (42)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral neuropathy (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (2) | 3 (3) | 1 (1) | 13 (15)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 4 (8) | 3 (6) | 3 (15) | 6 (9) | 3 (3) | 29 (75)
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 2 (3) | 1 (1) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (3) | 4 (6) | 2 (2) | 9 (13)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Nocturia
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Tachypnea
Rhinitis Infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shingles (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) — Skin lesion
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Skin and subcutaneous tissue disorders - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hernia repair
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (5)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (7) | 1 (2) | 2 (10) | 5 (9) | 2 (3) | 19 (42)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hyperviscosity
Vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — HHV6 Viremia
Vomiting (Gastrointestinal disorders) | 1 (2) | 3 (4) | 2 (2) | 1 (1) | 4 (6) | 0 (0) | 8 (13)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 7 (11)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT01054196/Prot_SAP_000.pdf